CLINICAL TRIAL: NCT02048007
Title: Evaluating Impact of Azithromycin Mass Drug Administrations on All-cause Mortality and Antibiotic Resistance: Morbidity Study
Brief Title: Mortality Reduction After Oral Azithromycin: Morbidity Study
Acronym: MORDORMorb
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPP1032340-B
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Childhood Mortality
Keywords: Childhood mortality; Azithromycin; Mass treatment; Infection; Bacterial infections; Trachoma; Chlamydia infections; Malaria; Diarrhea; Respiratory Infections; Antibiotic resistance; Verbal Autopsy; Microbiome
MeSH Terms: conditions — Infections; Bacterial Infections; Trachoma; Chlamydia Infections; Malaria; Diarrhea; Respiratory Tract Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biannual mass oral azithromycin (Active Comparator): Comparison of childhood infectious and nutritional morbidity in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months for 2 years
  Morbidity monitoring:
  Collect swabs (nasopharyngeal, nasal, conjunctival), blood samples, (thick/thin blood smears, hemoglobin, dried blood spots), and stool samples from 40 randomly selected children aged 1 month to 60 months per community; collect swabs (nasopharyngeal) from 40 randomly selected children aged 7-12 years per community.
  Anthropometry for all children aged 1 to 60 months per community.
  Collect nasopharyngeal swabs from all children aged 1-60 months who are seen at a local health clinic and have a respiratory complaint.
  Interventions: Drug: Azithromycin
- Biannual mass oral placebo (Placebo Comparator): Comparison of childhood infectious and nutritional morbidity in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo every 6 months for 2 years
  Collect swabs (nasopharyngeal, nasal, conjunctival), blood samples, (thick/thin blood smears, hemoglobin, dried blood spots), and stool samples from 40 randomly selected children aged 1 month to 60 months per community; collect swabs (nasopharyngeal) from 40 randomly selected children aged 7-12 years per community
  Anthropometry for all children aged 1 to 60 months per community
  Collect nasopharyngeal swabs from all children aged 1-60 months who are seen at a local health clinic and have a respiratory complaint
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Biannual mass oral azithromycin to children
  Other Names: Zithromax
  Arms: Biannual mass oral azithromycin
Drug: Placebo — Biannual mass oral placebo to children
  Arms: Biannual mass oral placebo

SUMMARY:
The long-term goal of this study is to more precisely define the role of mass azithromycin treatments as an intervention for reducing childhood morbidity and increasing growth, and for the potential selection of antibiotic resistance. The investigators propose a set of 3 cluster-randomized trials in Malawi, Niger, and Tanzania comparing communities randomized to oral azithromycin with those randomized to placebo. To assess the generalizability of the intervention, investigators will monitor for antibiotic resistance, which could potentially limit adoption of mass antibiotic treatments. The investigators will also assess several measures of infectious diseases. The investigators hypothesize that mass azithromycin treatments will reduce childhood morbidity and will be accompanied by an acceptable level of antibiotic resistance.

DETAILED DESCRIPTION:
The investigators will assess childhood infectious disease morbidity and macrolide resistance over two years, comparing communities where children aged 1-60 months receive biannual oral azithromycin to communities where the children receive biannual oral placebo.

Randomization of Treatment Allocation. In each site, 30 communities within a contiguous area of 300,000 to 600,000 individuals will be randomized into the azithromycin or placebo arm. The investigators will use a simple random sample separately for each study site, but without stratification or block randomization within the site. These communities are being randomized from the same pool of communities eligible for a sister trial (Mortality Reduction After Oral Azithromycin (MORDOR) - Morbidity Study).

Specific Aims

Specific Aim 1: To assess whether macrolide resistance is greater in a population-based community sample of pre-school children, or in a clinic-based sample of ill pre-school children

Specific Aim 2: To assess whether biannual mass azithromycin treatments of pre-school children can eliminate ocular chlamydia in a hypoendemic area

Specific Aim 3: To assess the diversity of the microbiome of the nasopharynx, nares, conjunctiva, and gastrointestinal tract

ELIGIBILITY:
Inclusion Criteria:

Communities:

* The community location in target district.
* The community leader consents to participation in the trial
* The community's estimated population is between 200-2,000 people.
* The community is not in an urban area.

Individuals (Intervention):

- Children-treated arms (all 3 sites): All children aged 1-60 months (up to but not including the 5th birthday), as assessed at the most recent biannual census

Individuals (Examination & Sample Collection):

* All swabs, blood tests, and stool samples: A random sample of children aged 1-60 months (up to but not including the 5th birthday) based on the previous census
* Anthropometric measurements: All children aged 1-60 months (up to but not including the 5th birthday) will have anthropometric measurements assessed.
* Nasopharyngeal swabs in untreated children: A random sample of individuals aged 7 - 12 years (7th birthday up to but not including the 12th birthday), as assessed from the previous census
* Clinic-based nasopharyngeal swabs: All children aged 1-60 months (up to but not including the 5th birthday) who present to a local health clinic in the study area and report symptoms of a respiratory infection

Exclusion Criteria:

Individuals:

* Pregnant women
* All those who are allergic to macrolides or azalides
* Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72000 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Presence of malaria parasites on thick blood smear or Rapid Diagnostic Test (RDT) in children 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Fraction of isolates of pneumococcus exhibiting macrolide resistance by nasopharyngeal swabs in children 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 36 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Prevalence of macrolide resistance in the stool as determined by genetic determinants or phenotypic testing | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Fraction of conjunctival swabs yielding ocular chlamydia in children 1-60 months | 24 months
  MORDOR Malawi and Niger. Please note: Each outcome will be analyzed separately for each study site.
Height over time in children aged 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi and Niger Please note: Each outcome will be analyzed separately in each of the two study sites.
Weight for Height over time in children aged 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi and Niger Please note:Each outcome will be analyzed separately in each of the two study sites.

SECONDARY OUTCOMES:
Density of asexual stages and gametocytes, in children 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi and Niger Please note: Each outcome will be analyzed separately in each of the two study sites.
Hemoglobin concentration and presence of anemia (hemoglobin <11 g/dL) in children 1-60 months | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Genetic determinants of macrolide resistance in the nasopharynx (eg pneumococcal) in individuals 7-12 years of age | 24 months
  MORDOR Niger
Genetic determinants of macrolide resistance in the nasopharynx (eg pneumococcal) in individuals 1-60 month olds seen in local health clinics for a respiratory complaint | 24 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Rates of acute respiratory illness among children 1-60 months. | 6-24 months after baseline
  MORDOR Tanzania
Presence of the trachoma grades "follicular trachoma" (TF) and "intense inflammatory trachoma" (TI), as defined by the World Health Organization (WHO) simplified grading system, in children 1-60 months | 24 months
  MORDOR Malawi and Niger Please note: Each outcome will be analyzed separately for each study site.
Rates of diarrhea among children (1-60 months) | 6-24 months after baseline
  MORDOR Tanzania
Proportion of rectal/stool isolates with evidence of resistance (in for example E.coli) to macrolides and other antibiotics commonly used to treat pediatric infections among children 1-60 months | 6-24 months after baseline; Niger will also report outcomes at 48 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Proportions of E. coli isolates resistant to macrolides and to antibiotics commonly used to treat pediatric infections among children 1-60 months hospitalized for pneumonia and diarrhea. | 6-24 months after baseline
  MORDOR Tanzania
Studies of intestinal permeability and inflammation, microbial translocation, and immune activation assessed through venous sampling of children 6 months | 5 x over 24 weeks after baseline
  MORDOR Malawi
Studies of intestinal permeability and inflammation, microbial translocation, and immune activation assessed through urine samples for L:M ratios of children 6 months | 5 x over 24 weeks after baseline
  MORDOR Malawi
Studies of intestinal permeability and inflammation, microbial translocation, and immune activation assessed through stool (fecal neopterin) of children 6 months | 5 x over 24 weeks after baseline
  MORDOR Malawi
Nasopharyngeal pneumococcal evidence of beta lactam and macrolide resistance in in children 1-60 months as measured by RNA-sequencing of the resistome | Tanzania will report outcomes at 6-24 months. Each site will report outcomes at 24 months; Niger will also report outcomes at 36 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Nasopharyngeal pneumococcal macrolide resistance determinants (eg erythromycin ribosomal methylase B and mefA), serotype, and multilocus sequence type in children 1-60 months | 24 months
  MORDOR Niger
Microbiome in the stool, nasopharynx, nares, and conjunctiva in children aged 1-59 months, as measured using next generation sequencing. Arms will be compared using Euclidean distance and diversity compared using Simpson's index. | 24 months
  Investigators will examine the effects of mass azithromycin (pre-treatment and post-treatment) on the human microbiome of African children by performing metagenomic experiments.
  MORDOR Niger
Microbial diversity in the intestinal microbiomes of children aged 1-60 months as measured by using next generation sequencing | 24 months
  Investigators will examine the effects of mass azithromycin (pre-treatment and post-treatment) on the human microbiome of African children by performing metagenomic experiments.
  MORDOR Malawi
Serology for exposure to exotic pathogens of children aged 1-60 months as measured by lateral flow assays or Multiplex bead array | 24 months
  MORDOR Malawi
Head circumference over time in children aged 1-60 months | 24 months
  MORDOR Malawi
Knee-heel length over time in children aged 1-60 months | 24 months
  MORDOR Malawi
Resistance (in E.coli phenotypically or genetic determinants) in stool of children aged 1-60 months. | Each site will report outcomes at 24 months; Niger will also report outcomes at 48 months
  MORDOR Malawi, Tanzania and Niger. Please note: Each outcome will be analyzed separately for each study site.
Prevalence of carriage of a panel of gastrointestinal parasites (Ancylostoma duodenale, Necator americanus, Ascaris lumbricoides, Trichuris trichiura, Giardia lamblia, Cryptosporidium hominis) of children aged 1-60 months | Baseline
  MORDOR Malawi
Prevalence of helicobacter pylori of children aged 1-60 months | Baseline
  MORDOR Malawi
Antibody response to enteric pathogens and malaria measured with a multiplex bead assay from dried blood spots collected from children 1 - 59 months | Niger will report outcomes at 36, 48 and 60 months
  MORDOR Niger

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Elodie J Lebas, RN, Study Director — University of California, San Francisco
Locations (6):
- United States (2):
  - UCSF Proctor Foundation, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
- College of Medicine at the University of Malawi, Blantyre, Blantyre, Malawi
- The Carter Center, Niger, Niamey, Niger
- Kongwa Trachoma Project, Kongwa, Tanzania
- London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arzika AM, Abdou A, Maliki R, Lebas E, Cook C, Vanderschelden B, O'Brien KS, Cotter SY, Varnado NE, Callahan EK, Bailey RL, West SK, Rosenthal PJ, Porco TC, Lietman TM, Keenan JD; MORDOR-Niger Study Group. Biannual Mass Azithromycin Distributions for Preschool Children and Malaria Parasitemia: A Secondary Analysis of the MORDOR Cluster Randomized Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2527148. doi: 10.1001/jamanetworkopen.2025.27148. PMID 40824641
- [Derived] Liu J, Brennhofer SA, Zhang J, Stroup S, Pholwat S, Arzika AM, Maliki R, Abdou A, Lebas E, O'Brien KS, Arnold BF, Keenan JD, Lietman TM, Platts-Mills JA, Rogawski McQuade ET, Houpt ER. Effect of biannual azithromycin on respiratory pathogens among symptomatic children: results from the randomised Macrolides Oraux pour Reduire les Deces avec un Oeil sur la Resistance (MORDOR) I trial. BMJ Glob Health. 2025 Feb 10;10(2):e016043. doi: 10.1136/bmjgh-2024-016043. PMID 39929535
- [Derived] Arzika AM, Mindo-Panusis D, Abdou A, Kadri B, Nassirou B, Maliki R, Alsoudi AF, Zhang T, Cotter SY, Lebas E, O'Brien KS, Callahan EK, Bailey RL, West SK, Goodhew EB, Martin DL, Arnold BF, Porco TC, Lietman TM, Keenan JD; Macrolides Oraux pour Reduire les Deces Avec un Oeil sur la Resistance (MORDOR)-Niger Study Group. Effect of Biannual Mass Azithromycin Distributions to Preschool-Aged Children on Trachoma Prevalence in Niger: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2228244. doi: 10.1001/jamanetworkopen.2022.28244. PMID 35997979
- [Derived] Arzika AM, Maliki R, Goodhew EB, Rogier E, Priest JW, Lebas E, O'Brien KS, Le V, Oldenburg CE, Doan T, Porco TC, Keenan JD, Lietman TM, Martin DL, Arnold BF; MORDOR-Niger Study Group. Effect of biannual azithromycin distribution on antibody responses to malaria, bacterial, and protozoan pathogens in Niger. Nat Commun. 2022 Feb 21;13(1):976. doi: 10.1038/s41467-022-28565-5. PMID 35190534
- [Derived] Hart JD, Samikwa L, Meleke H, Burr SE, Cornick J, Kalua K, Bailey RL. Prevalence of nasopharyngeal Streptococcus pneumoniae carriage and resistance to macrolides in the setting of azithromycin mass drug administration: analysis from a cluster-randomised controlled trial in Malawi, 2015-17. Lancet Microbe. 2022 Feb;3(2):e142-e150. doi: 10.1016/S2666-5247(21)00279-2. PMID 35156069
- [Derived] Arzika AM, Maliki R, Ali MM, Alio MK, Abdou A, Cotter SY, Varnado NE, Lebas E, Cook C, Oldenburg CE, O'Brien KS, Callahan EK, Bailey RL, West SK, Porco TC, Lietman TM, Keenan JD; MORDOR-Niger Study Group. Effect of Mass Azithromycin Distributions on Childhood Growth in Niger: A Cluster-Randomized Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2139351. doi: 10.1001/jamanetworkopen.2021.39351. PMID 34967883
- [Derived] Bloch EM, Mrango Z, Weaver J, Munoz B, Lietman TM, West SK. Causes of death after biannual azithromycin treatment: A community-level randomized clinical trial. PLoS One. 2021 Sep 24;16(9):e0250197. doi: 10.1371/journal.pone.0250197. eCollection 2021. PMID 34559801
- [Derived] Arzika AM, Maliki R, Boubacar N, Kane S, Cotter SY, Lebas E, Cook C, Bailey RL, West SK, Rosenthal PJ, Porco TC, Lietman TM, Keenan JD; MORDOR Study Group. Biannual mass azithromycin distributions and malaria parasitemia in pre-school children in Niger: A cluster-randomized, placebo-controlled trial. PLoS Med. 2019 Jun 25;16(6):e1002835. doi: 10.1371/journal.pmed.1002835. eCollection 2019 Jun. PMID 31237871
- [Derived] West SK, Bloch E, Weaver J, Munoz B, Mrango Z, Kasubi M, Lietman T, Coles C. Morbidity in a Longitudinal Cohort of Children Residing in Villages Randomized to Biannual Treatment With Azithromycin Versus Placebo. Clin Infect Dis. 2020 Feb 3;70(4):574-580. doi: 10.1093/cid/ciz269. PMID 30950493
- [Derived] Oldenburg CE, Arzika AM, Maliki R, Kane MS, Lebas E, Ray KJ, Cook C, Cotter SY, Zhou Z, West SK, Bailey R, Porco TC, Keenan JD, Lietman TM; MORDOR Study Group. Safety of azithromycin in infants under six months of age in Niger: A community randomized trial. PLoS Negl Trop Dis. 2018 Nov 12;12(11):e0006950. doi: 10.1371/journal.pntd.0006950. eCollection 2018 Nov. PMID 30419040
- [Derived] Doan T, Hinterwirth A, Arzika AM, Cotter SY, Ray KJ, O'Brien KS, Zhong L, Chow ED, Zhou Z, Cummings SL, Fry D, Oldenburg CE, Worden L, Porco TC, Keenan JD, Lietman TM. Mass Azithromycin Distribution and Community Microbiome: A Cluster-Randomized Trial. Open Forum Infect Dis. 2018 Jul 24;5(8):ofy182. doi: 10.1093/ofid/ofy182. eCollection 2018 Aug. PMID 30151409
- [Derived] Doan T, Arzika AM, Ray KJ, Cotter SY, Kim J, Maliki R, Zhong L, Zhou Z, Porco TC, Vanderschelden B, Keenan JD, Lietman TM. Gut Microbial Diversity in Antibiotic-Naive Children After Systemic Antibiotic Exposure: A Randomized Controlled Trial. Clin Infect Dis. 2017 May 1;64(9):1147-1153. doi: 10.1093/cid/cix141. PMID 28402408
- [Derived] Porco TC, Stoller NE, Keenan JD, Bailey RL, Lietman TM. Public key cryptography for quality assurance in randomization for clinical trials. Contemp Clin Trials. 2015 May;42:167-8. doi: 10.1016/j.cct.2015.03.016. Epub 2015 Apr 7. No abstract available. PMID 25858004